CLINICAL TRIAL: NCT00810732
Title: THE EFFECTS OF SITAXSENTAN ONCE DAILY DOSING ON PROTEINURIA, 24-HOUR BLOOD PRESSURE, AND ARTERIAL STIFFNESS IN SUBJECTS WITH CHRONIC KIDNEY DISEASE
Brief Title: Effects Of Sitaxsentan On Proteinuria, 24-Hour Blood Pressure, And Arterial Stiffness In Chronic Kidney Disease Subjects
Acronym: FCRD01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B1321005; B1321005; 2006-002004-33 (EudraCT Number); FCRD01 (Other: Alias Study Number)
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Results first posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2022-08

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Sitaxsentan
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — sitaxsentan; Nifedipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sitaxsentan (Experimental): Sitaxsentan sodium 100 mg orally administered once daily (double blind arm)
  Interventions: Drug: Open
- Nifedipine (Active Comparator): Nifedipine 30 mg extended release tablets, orally administered once daily (open label arm)
  Interventions: Drug: Nifedipine
- Placebo (Placebo Comparator): Placebo for sitaxsentan, orally administered once daily (double blind arm)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Open — Sitaxsentan sodium 100 mg orally administered once daily (double blind arm)
  Other Names: Sitaxsentan
  Arms: Sitaxsentan
Drug: Nifedipine — Nifedipine = 30 mg extended release tablets, orally administered once daily (open label arm)
  Arms: Nifedipine
Drug: Placebo — Placebo for sitaxsentan, orally administered once daily (double blind arm)
  Arms: Placebo

SUMMARY:
This study is being conducted to evaluate sitaxsentan dosing in subjects with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Has stage 1-5 chronic kidney disease (CKD) as defined by the Kidney Disease Outcomes Quality Initiative (K/DOQI) with proteinuria, including any of the following aetiologies: immunoglobulin (IgA) nephropathy, polycystic kidney disease (PCKD), congenital abnormalities, reflux nephropathy, focal segmental glomerulosclerosis, minimal change nephropathy, and membranous nephropathy.

Exclusion Criteria:

* Required peritoneal dialysis or haemodialysis.
* Has kidney disease due to diabetes mellitus, vasculitis, systemic lupus erythematosus, or known renovascular disease; antiglomerular basement membrane disease; or is on immunosuppressive medication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-05-09 (Actual); Primary Completion 2009-03-06 (Actual); Study Completion 2009-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United Kingdom (2):
  - Clinical Research Centre and Pharmacology Unit, Edinburgh, Scotland
  - the University of Edinburgh, Western General Hospital, Department of Medical Sciences, Edinburgh, Scotland

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Farrah TE, Anand A, Gallacher PJ, Kimmitt R, Carter E, Dear JW, Mills NL, Webb DJ, Dhaun N. Endothelin Receptor Antagonism Improves Lipid Profiles and Lowers PCSK9 (Proprotein Convertase Subtilisin/Kexin Type 9) in Patients With Chronic Kidney Disease. Hypertension. 2019 Aug;74(2):323-330. doi: 10.1161/HYPERTENSIONAHA.119.12919. Epub 2019 Jun 10. PMID 31177906
- [Derived] Dhaun N, Yuzugulen J, Kimmitt RA, Wood EG, Chariyavilaskul P, MacIntyre IM, Goddard J, Webb DJ, Corder R. Plasma pro-endothelin-1 peptide concentrations rise in chronic kidney disease and following selective endothelin A receptor antagonism. J Am Heart Assoc. 2015 Mar 23;4(3):e001624. doi: 10.1161/JAHA.114.001624. PMID 25801761
- [Derived] Dhaun N, Moorhouse R, MacIntyre IM, Melville V, Oosthuyzen W, Kimmitt RA, Brown KE, Kennedy ED, Goddard J, Webb DJ. Diurnal variation in blood pressure and arterial stiffness in chronic kidney disease: the role of endothelin-1. Hypertension. 2014 Aug;64(2):296-304. doi: 10.1161/HYPERTENSIONAHA.114.03533. PMID 24890823
- [Derived] Dhaun N, Melville V, Blackwell S, Talwar DK, Johnston NR, Goddard J, Webb DJ. Endothelin-A receptor antagonism modifies cardiovascular risk factors in CKD. J Am Soc Nephrol. 2013 Jan;24(1):31-6. doi: 10.1681/ASN.2012040355. Epub 2012 Dec 14. PMID 23243212
- [Derived] Dhaun N, MacIntyre IM, Kerr D, Melville V, Johnston NR, Haughie S, Goddard J, Webb DJ. Selective endothelin-A receptor antagonism reduces proteinuria, blood pressure, and arterial stiffness in chronic proteinuric kidney disease. Hypertension. 2011 Apr;57(4):772-9. doi: 10.1161/HYPERTENSIONAHA.110.167486. Epub 2011 Feb 28. PMID 21357275
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1321005&StudyName=Effects%20Of%20Sitaxsentan%20On%20Proteinuria%2C%2024-Hour%20Blood%20Pressure%2C%20And%20Arterial%20Stiffness%20In%20Chronic%20Kidney%20Disease%20Subjects

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then Sitaxsentan Then Nifedipine: Participants received placebo matched to Sitaxsentan 100 milligram (mg) tablet orally, once daily for 6 weeks in first intervention period, then Sitaxsentan 100 mg tablet orally, once daily for 6 weeks in second intervention period, followed by Nifedipine extended release (ER) 30 mg tablet orally, once daily for 6 weeks in third intervention period. Each intervention period was separated by a washout period of at least 2 weeks.
- Sitaxsentan Then Nifedipine Then Placebo: Participants received Sitaxsentan 100 mg tablet orally, once daily for 6 weeks in first intervention period, then nifedipine ER 30 mg tablet orally, once daily for 6 weeks in second intervention period, followed by placebo matched Sitaxsentan 100 mg tablet orally, once daily for 6 weeks in third intervention period. Each intervention period was separated by a washout period of at least 2 weeks.
- Nifedipine Then Sitaxsentan Then Placebo: Participants received Nifedipine ER 30 mg tablet orally, once daily for 6 weeks in first intervention period, then Sitaxsentan 100 mg tablet orally, once daily for 6 weeks in second intervention period, followed by placebo matched to Sitaxsentan 100 mg tablet orally, once daily for 6 weeks in third intervention period. Each intervention period was separated by a washout period of at least 2 weeks.
- Nifedipine Then Placebo Then Sitaxsentan: Participants received Nifedipine ER 30 mg tablet orally, once daily for 6 weeks in first intervention period, then placebo matched to Sitaxsentan 100 mg tablet orally, once daily for 6 weeks in second intervention period, followed by Sitaxsentan 100 mg tablet orally, once daily for 6 weeks in third intervention period. Each intervention period was separated by a washout period of at least 2 weeks.
- Placebo Then Nifedipine Then Sitaxsentan: Participants received placebo matched to Sitaxsentan 100 mg tablet orally, once daily for 6 weeks in first intervention period, then Nifedipine ER 30 mg tablet orally, once daily for 6 weeks in second intervention period, followed by Sitaxsentan 100 mg tablet orally, once daily for 6 weeks in third intervention period. Each intervention period was separated by a washout period of at least 2 weeks.
- Sitaxsentan Then Placebo Then Nifedipine: Participants received Sitaxsentan 100 mg tablet orally, once daily for 6 weeks in first intervention period, then placebo matched to Sitaxsentan 100 mg tablet orally, once daily for 6 weeks in second intervention period, followed by Nifedipine ER 30 mg tablet orally, once daily for 6 weeks in third intervention period. Each intervention period was separated by a washout period of at least 2 weeks.
Period: First Intervention Period (6 Weeks)
Arm/Group | Placebo Then Sitaxsentan Then Nifedipine | Sitaxsentan Then Nifedipine Then Placebo | Nifedipine Then Sitaxsentan Then Placebo | Nifedipine Then Placebo Then Sitaxsentan | Placebo Then Nifedipine Then Sitaxsentan | Sitaxsentan Then Placebo Then Nifedipine
Started | 5 | 4 | 4 | 5 | 5 | 4
Completed | 5 | 4 | 4 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: First Washout Period (at Least 2 Weeks)
Arm/Group | Placebo Then Sitaxsentan Then Nifedipine | Sitaxsentan Then Nifedipine Then Placebo | Nifedipine Then Sitaxsentan Then Placebo | Nifedipine Then Placebo Then Sitaxsentan | Placebo Then Nifedipine Then Sitaxsentan | Sitaxsentan Then Placebo Then Nifedipine
Started | 5 | 4 | 4 | 5 | 5 | 4
Completed | 5 | 4 | 4 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention Period (6 Weeks)
Arm/Group | Placebo Then Sitaxsentan Then Nifedipine | Sitaxsentan Then Nifedipine Then Placebo | Nifedipine Then Sitaxsentan Then Placebo | Nifedipine Then Placebo Then Sitaxsentan | Placebo Then Nifedipine Then Sitaxsentan | Sitaxsentan Then Placebo Then Nifedipine
Started | 5 | 4 | 4 | 5 | 5 | 4
Completed | 5 | 4 | 4 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Washout Period (at Least 2 Weeks)
Arm/Group | Placebo Then Sitaxsentan Then Nifedipine | Sitaxsentan Then Nifedipine Then Placebo | Nifedipine Then Sitaxsentan Then Placebo | Nifedipine Then Placebo Then Sitaxsentan | Placebo Then Nifedipine Then Sitaxsentan | Sitaxsentan Then Placebo Then Nifedipine
Started | 5 | 4 | 4 | 5 | 5 | 4
Completed | 5 | 4 | 4 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention Period (6 Weeks)
Arm/Group | Placebo Then Sitaxsentan Then Nifedipine | Sitaxsentan Then Nifedipine Then Placebo | Nifedipine Then Sitaxsentan Then Placebo | Nifedipine Then Placebo Then Sitaxsentan | Placebo Then Nifedipine Then Sitaxsentan | Sitaxsentan Then Placebo Then Nifedipine
Started | 5 | 4 | 4 | 5 | 5 | 4
Completed | 5 | 4 | 4 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who received at least one dose of study drug and had received at least 1 on-treatment assessment for at least 1 endpoint.
Groups:
- Overall Study: All participants who were randomized to receive Sitaxsentan 100 mg tablet, Nifedipine ER 30 mg tablet and placebo matched to Sitaxsentan 100 mg tablet orally, once daily for 6 weeks in any intervention period. Each intervention period was separated by a washout period of at least 2 weeks.
Arm/Group | Overall Study
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean 24-Hour Urine Total Protein Level at Week 6
Description: Mean urine total protein assessment included 24-hour urine collections to assess total protein excretion per 24 hours. Baseline was derived from an average of Week 0 (pre-dose) 24-hour urine collections prior to each treatment period. Week 6 was derived from an average of Week 6 24-hour urine collections for each treatment period.
Time Frame: Baseline, Week 6
Population: FAS included all participants who received at least one dose of study drug and had received at least 1 on-treatment assessment for at least 1 endpoint.
Measure: Mean (Standard Deviation); unit: Grams per 24 hours
Groups:
- Sitaxsentan: Participants received Sitaxsentan 100 mg tablet orally, once daily for 6 weeks in either first, second or third intervention period.
- Placebo: Participants administered placebo matched to 100 mg tablets orally, once daily for 6 weeks in either first, second or third intervention period.
- Nifedipine: Participants were administered Nifedipine 30 mg ER tablet orally, once daily for 6 weeks in either first, second or third intervention period.
Arm/Group | Sitaxsentan | Placebo | Nifedipine
Number analyzed (Participants) | 27 | 27 | 27
Grams per 24 hours
  Baseline | 2.07 (1.77) | 2.07 (1.96) | 1.95 (1.58)
  Change at week 6 | -0.62 (0.56) | -0.06 (0.89) | 0.01 (0.77)
Statistical Analysis 1: Comparison: Sitaxsentan vs Placebo; Test type: Superiority or Other; p = 0.0040, ANCOVA; Least Squares (LS) Mean Difference = -0.56, 95% CI 2-sided [-0.94 to -0.19], Standard Error of Mean 0.19
Statistical Analysis 2: Comparison: Sitaxsentan vs Nifedipine; Test type: Superiority or Other; p = 0.0018, ANCOVA; LS Mean Difference = -0.61, 95% CI 2-sided [-0.99 to -0.24], Standard Error of Mean 0.19
Statistical Analysis 3: Comparison: Placebo vs Nifedipine; Test type: Superiority or Other; p = 0.7945, ANCOVA; LS Mean Difference = 0.05, 95% CI 2-sided [-0.33 to 0.43], Standard Error of Mean 0.19

2. Secondary Outcome: Change From Baseline in Mean Systemic Arterial Blood Pressure (BP), Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Week 3 and 6
Description: The 24-hour ambulatory BP monitoring was performed by using a BP cuff which was attached to the participant's arm, using the same arm throughout the study, with a small monitor that comfortably sits in the pocket of participant. Mean values over 24-hour measurements at each measurement period were calculated. The change in total 24-hour ambulatory monitoring of systemic arterial BP, SBP and DBP at Week 3 and 6 relative to baseline were reported. Baseline was as an average of the pre-dose measurement for the measure collected at Week 0 of each treatment period. Week 3 and Week 6 was an average of measurement for the measure collected at Week 3 and 6 of each treatment period.
Time Frame: Baseline, Week 3 and 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeter of Mercury (mmHg)
Arm/Group | Sitaxsentan | Placebo | Nifedipine
Number analyzed (Participants) | 27 | 27 | 27
Millimeter of Mercury (mmHg)
  Mean Systemic Arterial BP: Baseline | 92.94 (7.39) | 92.98 (9.33) | 93.78 (8.35)
  Mean Systemic Arterial BP: Change at Week 3 | -4.59 (5.02) | -1.20 (4.70) | -2.95 (5.90)
  Mean Systemic Arterial BP: Change at Week 6 | -3.74 (5.62) | -0.35 (5.38) | -3.54 (5.49)
  Mean Systemic Arterial SBP :Baseline | 124.03 (11.44) | 125.17 (13.95) | 125.12 (12.33)
  Mean Systemic Arterial SBP: Change at Week 3 | -4.88 (7.34) | -2.81 (7.21) | -4.20 (7.67)
  Mean Systemic Arterial SBP: Change at Week 6 | -3.99 (7.82) | -1.57 (7.22) | -4.47 (7.97)
  Mean Systemic Arterial DBP: Baseline | 77.56 (6.67) | 77.58 (8.05) | 78.27 (7.74)
  Mean Systemic Arterial DBP: Change at Week 3 | -4.85 (4.51) | -0.86 (3.98) | -2.09 (5.59)
  Mean Systemic Arterial DBP: Change at Week 6 | -3.60 (5.02) | -0.41 (5.03) | -2.86 (4.92)
Statistical Analysis 1: Comparison: Sitaxsentan vs Placebo; Mean Systemic Arterial BP: Week 3; Test type: Superiority or Other; p = 0.0087, ANCOVA; LS mean difference = -3.50, 95% CI 2-sided [-6.08 to -0.91], Standard Error of Mean 1.30
Statistical Analysis 2: Comparison: Sitaxsentan vs Nifedipine; Mean Systemic Arterial BP: Week 3; Test type: Superiority or Other; p = 0.1424, ANCOVA; LS mean difference = -1.92, 95% CI 2-sided [-4.50 to 0.66], Standard Error of Mean 1.30
Statistical Analysis 3: Comparison: Placebo vs Nifedipine; Mean Systemic Arterial BP: Week 3; Test type: Superiority or Other; p = 0.2277, ANCOVA; LS mean difference = -1.58, 95% CI 2-sided [-4.15 to 1.00], Standard Error of Mean 1.29
Statistical Analysis 4: Comparison: Sitaxsentan vs Placebo; Systolic Blood Pressure: Week 3; Test type: Superiority or Other; p = 0.1599, ANCOVA; LS mean difference = -2.56, 95% CI 2-sided [-6.16 to 1.03], Standard Error of Mean 1.81
Statistical Analysis 5: Comparison: Sitaxsentan vs Nifedipine; Systolic Blood Pressure: Week 3; Test type: Superiority or Other; p = 0.5545, ANCOVA; LS mean difference = -1.07, 95% CI 2-sided [-4.66 to 2.52], Standard Error of Mean 1.80
Statistical Analysis 6: Comparison: Placebo vs Nifedipine; Systolic Blood Pressure: Week 3; Test type: Superiority or Other; p = 0.4095, ANCOVA; LS mean difference = -1.49, 95% CI 2-sided [-5.08 to 2.09], Standard Error of Mean 1.80
Statistical Analysis 7: Comparison: Sitaxsentan vs Placebo; Diastolic Blood Pressure: Week 3; Test type: Superiority or Other; p = 0.0012, ANCOVA; LS mean difference = -4.08, 95% CI 2-sided [-6.49 to -1.67], Standard Error of Mean 1.21
Statistical Analysis 8: Comparison: Sitaxsentan vs Nifedipine; Diastolic Blood Pressure: Week 3; Test type: Superiority or Other; p = 0.0159, ANCOVA; LS mean difference = -2.98, 95% CI 2-sided [-5.38 to -0.57], Standard Error of Mean 1.21
Statistical Analysis 9: Comparison: Placebo vs Nifedipine; Diastolic Blood Pressure: Week 3; Test type: Superiority or Other; p = 0.3627, ANCOVA; LS mean difference = -1.10, 95% CI 2-sided [-3.51 to 1.30], Standard Error of Mean 1.21
Statistical Analysis 10: Comparison: Sitaxsentan vs Placebo; Mean Systemic Arterial BP: Week 6; Test type: Superiority or Other; p = 0.0057, ANCOVA; LS mean difference = -3.36, 95% CI 2-sided [-5.69 to -1.03], Standard Error of Mean 1.16
Statistical Analysis 11: Comparison: Sitaxsentan vs Nifedipine; Mean Systemic Arterial BP: Week 6; Test type: Superiority or Other; p = 0.6503, ANCOVA; LS mean difference = -0.53, 95% CI 2-sided [-2.86 to 1.80], Standard Error of Mean 1.16
Statistical Analysis 12: Comparison: Placebo vs Nifedipine; Mean Systemic Arterial BP: Week 6; Test type: Superiority or Other; p = 0.0183, ANCOVA; LS mean difference = -2.83, 95% CI 2-sided [-5.16 to -0.50], Standard Error of Mean 1.16
Statistical Analysis 13: Comparison: Sitaxsentan vs Placebo; Systolic Blood Pressure (SBP): Week 6; Test type: Superiority or Other; p = 0.0726, ANCOVA; LS mean difference = -2.81, 95% CI 2-sided [-5.89 to 0.27], Standard Error of Mean 1.53
Statistical Analysis 14: Comparison: Sitaxsentan vs Nifedipine; Systolic Blood Pressure (SBP): Week 6; Test type: Superiority or Other; p = 0.9661, ANCOVA; LS mean difference = 0.07, 95% CI 2-sided [-3.01 to 3.14], Standard Error of Mean 1.53
Statistical Analysis 15: Comparison: Placebo vs Nifedipine; Systolic Blood Pressure (SBP): Week 6; Test type: Superiority or Other; p = 0.0656, ANCOVA; LS mean difference = -2.88, 95% CI 2-sided [-5.94 to 0.19], Standard Error of Mean 1.53
Statistical Analysis 16: Comparison: Sitaxsentan vs Placebo; Diastolic Blood Pressure (DBP): Week 6; Test type: Superiority or Other; p = 0.0068, ANCOVA; LS mean difference = -3.16, 95% CI 2-sided [-5.39 to -0.92], Standard Error of Mean 1.11
Statistical Analysis 17: Comparison: Sitaxsentan vs Nifedipine; Diastolic Blood Pressure (DBP): Week 6; Test type: Superiority or Other; p = 0.3760, ANCOVA; LS mean difference = -0.99, 95% CI 2-sided [-3.22 to 1.24], Standard Error of Mean 1.11
Statistical Analysis 18: Comparison: Placebo vs Nifedipine; Diastolic Blood Pressure (DBP): Week 6; Test type: Superiority or Other; p = 0.0572, ANCOVA; LS mean difference = -2.16, 95% CI 2-sided [-4.40 to 0.07], Standard Error of Mean 1.11

3. Secondary Outcome: Change From Baseline in Carotid-Femoral Pulse Wave Velocity (PWV) at Week 3 and 6
Description: Carotid-femoral pulse wave velocity (PWV), a measure of arterial stiffness, is determined from the time taken for the arterial pulse to propagate from the carotid to the femoral artery. Baseline was defined as the pre-dose measurement for the measure collected at Week 0 of each treatment period. Week 3 and Week 6 was an average of measurement for the measure collected at Week 3 and 6 of each treatment period.
Time Frame: Baseline, Week 3 and 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Meter per second
Arm/Group | Sitaxsentan | Placebo | Nifedipine
Number analyzed (Participants) | 27 | 27 | 27
Meter per second
  Baseline | 7.97 (1.58) | 7.74 (1.58) | 7.94 (1.74)
  Change at Week 3 | -0.19 (0.95) | -0.21 (0.69) | -0.21 (0.92)
  Change at Week 6 | -0.41 (0.82) | 0.29 (1.08) | -0.38 (0.86)
Statistical Analysis 1: Comparison: Sitaxsentan vs Placebo; Week 3; Test type: Superiority or Other; p = 0.8823, ANCOVA; LS mean difference = 0.03, 95% CI 2-sided [-0.39 to 0.45], Standard Error of Mean 0.21
Statistical Analysis 2: Comparison: Sitaxsentan vs Nifedipine; Week 3; Test type: Superiority or Other; p = 0.9457, ANCOVA; LS mean difference = 0.01, 95% CI 2-sided [-0.41 to 0.43], Standard Error of Mean 0.21
Statistical Analysis 3: Comparison: Placebo vs Nifedipine; Week 3; Test type: Superiority or Other; p = 0.9358, ANCOVA; LS mean difference = 0.02, 95% CI 2-sided [-0.40 to 0.44], Standard Error of Mean 0.21
Statistical Analysis 4: Comparison: Sitaxsentan vs Placebo; Week 6; Test type: Superiority or Other; p = 0.0022, ANCOVA; LS mean difference = -0.64, 95% CI 2-sided [-1.03 to -0.25], Standard Error of Mean 0.19
Statistical Analysis 5: Comparison: Sitaxsentan vs Nifedipine; Week 6; Test type: Superiority or Other; p = 0.8956, ANCOVA; LS mean difference = -0.03, 95% CI 2-sided [-0.41 to 0.36], Standard Error of Mean 0.19
Statistical Analysis 6: Comparison: Placebo vs Nifedipine; Week 6; Test type: Superiority or Other; p = 0.0030, ANCOVA; LS mean difference = -0.61, 95% CI 2-sided [-1.00 to -0.23], Standard Error of Mean 0.19

ADVERSE EVENTS:
Arm/Group | Sitaxsentan | Placebo | Nifedipine
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 13/27 | 21/27 | 18/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitaxsentan (N=27) | Placebo (N=27) | Nifedipine (N=27)
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 1
Eye disorder (Eye disorders) | 0 | 0 | 1
Iritis (Eye disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1
Fatigue (General disorders) | 1 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0
Balanitis candida (Infections and infestations) | 0 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Infusion site infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 3
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Dizziness (Nervous system disorders) | 1 | 2 | 1
Headache (Nervous system disorders) | 2 | 10 | 10
Migraine (Nervous system disorders) | 1 | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.